CLINICAL TRIAL: NCT06505772
Title: Dexmedetomidine Improves Oxygenation and Reduces Pulmonary Shunt in High-Risk Pediatric Patients Undergoing One-Lung Ventilation for Thoracic Surgery: A Double-Blind Randomized Controlled Trial at Damascus University Children's Hospital
Brief Title: Dexmedetomidine Improved Oxygenation and Reduced Shunt in One-Lung Ventilation at High-Risk Pediatric Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Collaborators: University Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UDMS-Anesth-02-2024
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: One-Lung Ventilation; Thoracic Surgery
Keywords: Hypoventilation pulmonary vasoconstriction HPV; Pulmonary shunt fraction Qs/Qt; Dexmedetomidine; partial pressure of arterial oxygen (PaO2)
MeSH Terms: interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Anesthesiologists, graduate students, anesthesiologists, patients and their families will not know if a child is taking the drug or not.
  Also, the person who will conduct the survey will not know either, all will be hidden.
  Depending on the volume in ml, to mask the medical team from the substance of the drug...
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The dexmedetomidine group (Experimental): Dexmedetomidine:
  An initial dose of 0.5 mcg/kg of dexmedetomidine will be given over 10 minutes, starting 10 minutes after the initiation of anesthesia infusion.
  Following the initial dose, a continuous infusion of dexmedetomidine will be administered at a rate of 0.4 mcg/kg/hour.
  The infusion will be stopped before skin closure.
  Interventions: Drug: Dexmedetomidine
- The Placebo group (the control group): (Placebo Comparator): Saline Solution (Placebo):
  After the induction of anesthesia, a volume of saline solution equivalent to the volume of dexmedetomidine used in the experimental group will be administered using the same protocol.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dexmedetomidine — Infusion syringes are supplied with a concentration of 0.25 mcg / mL (dexmedetomidine ) either 80 mcg / 20 mL, 200 mcg / 50 mL, or 400 mcg / 100 mL.
  For example, it begins with an infusion of 4 ml over 10 minutes and then continues the infusion, depending on the weight of the child, at a rate of 1.6 ml/kg/hour.
  All injections will be prepared randomly by a doctor who did not participate in the study, and then placed in unmarked infusion pumps, given to an anesthesiologist (more than 10 years experience in pediatric anesthesia) without knowledge of the infusion content. The randomization process is carried out via sealed envelope technique.
  The injections in both groups will be stopped before the skin is closed. Both patients and anesthesiologists blinded the study drug (dexmedetomidine or placebo) by infusion of solution (dexmedetomidine or placebo). Depending on the size in ml, to ensure that there is no bias and blindness to the medical team about what the drug is.
  Other Names: Precedex
  Arms: The dexmedetomidine group
Drug: Normal saline — Normal saline (NS) for intravenous infusion is supplied in pre-filled syringes of 20 ml, 50 ml, and 100 ml. To maintain blinding in this study, NS is handled identically to the study drug, dexmedetomidine. A physician not involved in the study prepares all injections, randomly assigning either NS or dexmedetomidine using a sealed envelope technique. Prepared syringes are then placed in identical, unmarked infusion pumps.
  Infusion Protocol:
  Anesthesiologists, blinded to the infusion contents, administer the solutions according to the protocol:
  For example,Initial Bolus: 4 ml infused over 10 minutes, Maintenance Infusion: Continued at a rate of 1.6 ml/kg/hour, adjusted to the individual patient's weight.
  This process ensures both patient and anesthesiologist remain blinded to the treatment arm, minimizing potential bias throughout the study.
  Other Names: Placebo
  Arms: The Placebo group (the control group):

SUMMARY:
Children with high anesthetic risk who underwent Thoracic surgery with OLV (one lung ventilation) technique during general anesthesia were divided into two groups.

The first is an intravenous injection of dexmedetomidine at a rate of 0.4 micrograms/kg/hour as a continuous intravenous infusion. The second group, the placebo group, injected the second with a normal saline solution, an infusion that will pass through the vein, using blinded, unmarked syringes.

Three arterial blood gas (ABG) samples were taken during surgery at designated times. Circulatory PaO2 values were recorded and the Qs/Qt shunt value was calculated.

DETAILED DESCRIPTION:
Pediatric specific anatomy and physiology includes small ventricles with low systolic mass and poor ventricular compliance . With decreased peripheral vascular resistance (SVR) . The parasympathetic nervous system is dominant. This explains why HR is delayed compared to changes in MAP and mean blood pressure, is less affected and slower to respond. As each terminal bronchiole opens into a single alveolus and initially forms clusters of clusters, rather than fully developed alveolar clusters, these clusters continue to grow until six to eight years of age to resemble adults. The diaphragm is more horizontal, which reduces its mechanical advantage. Ventilation depends mainly on the diaphragm and the rate of its movements (breathing movements). Higher compliance of the thoracic wall is also seen with increased respiratory work.

Decreased functional residual capacity (FRC) increases pulmonary shunting and leads to atelectasis. One-lung ventilation (OLV) during general anesthesia can improve the surgical field of view, which is often used in thoracic surgery. However, OLV can lead to a mismatch in the ventilation/perfusion ratio (V/Q), leading to increased shunt and pulmonary shunt fraction (Qs/Qt) within the lungs and the occurrence of hypoxia. The ratio between the rate of flow of unoxygenated blood from the pulmonary arteries to the pulmonary veins through the shunt (Qs), and the total rate of blood flow through the lungs (Qt), i.e., the ratio between the unoxygenated blood and the total blood, is known as the pulmonary shunt fraction (Qs/Qt). The FEV1/FVC ratio represents the proportion of the total vital capacity that can be exhaled in the first second of forced expiration, whereas FEV1 indicates "Force Expiratory Volume in 1 second" and FVC indicates "Forced Vital Capacity".

Hypoventilation-induced vasoconstriction (HPV) is the body's primary compensatory mechanism against pulmonary constriction, which is to divert pulmonary perfusion blood from the nonventilated area to the ventilated area, thereby reducing pulmonary constriction and improving blood hypoxia . HPV is affected by various factors, including changes in pulmonary pressure, alkalosis, vasodilators, and inhaled anesthetic gases, which have the greatest effect. The study was designed as a two-group, controlled clinical trial using propofol, which is known to have no effect on HPV.

Dexmedetomidine is widely used as an anesthetic adjuvant. It is a highly selective alpha2 adrenergic receptor agonist that directly stimulates peripheral alpha2 receptors to induce vasoconstriction and increase blood pressure, as well as act on central alpha2 receptors to suppress sympathetic excitation, which can dilate blood vessels and lower blood pressure. Alpha adrenal blockade eliminates pulmonary arrhythmias that responded to non-adrenal but not hypoxia . Due to the complex effects of dexmedetomidine on blood circulation, it is difficult to predict its effects on intrapulmonary shunt and hypoventilation-induced vasoconstriction in patients during one-lung ventilation . The hypothesis of our study predicted that dexmedetomidine would improve oxygenation Partial Pressure of Arterial Oxygen (PaO2) and reduce pulmonary shunting during OLV in children.

ELIGIBILITY:
Inclusion Criteria:

* children with American Society of Anesthesiologists (ASA) grade III
* FEV1/FVC values less than 80% . FEV1/FVC ratio represents the proportion of the total vital capacity that can be exhaled in the first second of forced expiration, whereas FEV1 indicates "Force Expiratory Volume in 1 second" and FVC indicates "Forced Vital Capacity".
* Qs/Qt ratio greater than 10 .

Exclusion Criteria:

* renal failure.
* hepatic dysfunction.
* congenital and valvular cardiac disease.
* neurological illnesses.
* During surgery, individuals who did not achieve complete lung isolation were excluded.
* During surgery, individuals with poor oxygen saturation (SO2 <90%) who did not react to maneuvers and anesthetic procedures to boost saturation were removed.
* During surgery, Participants who had a heart rate of less than 80 beats per minute, did not react to atropine, or required a dosage of inotropic drugs (dopamine) were also removed from the trial.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Change in the PaO2 | four time points: (T1) 10 minutes after initiation of total lung ventilation (TLV), (T2) 10 minutes after initiation of one-lung ventilation (OLV), (T3) 60 minutes after initiation of OLV, and (T4) 20 minutes after the end of OLV.
  Evaluation of Change in PaO2 During Surgery. PaO2: is Partial Pressure of Arterial Oxygen.
Change in the Qs/Qt | four time points: (T1) 10 minutes after initiation of total lung ventilation (TLV), (T2) 10 minutes after initiation of one-lung ventilation (OLV), (T3) 60 minutes after initiation of OLV, and (T4) 20 minutes after the end of OLV.
  Evaluation of Change in Qs/Qt During Surgery. Qs/Qt: is a Measurement of Pulmonary Shunt. Qs: Blood Flow Through the Shunt, Qt : Total Blood Flow.

SECONDARY OUTCOMES:
Change in the PIP | four time points: (T1) 10 minutes after initiation of total lung ventilation (TLV), (T2) 10 minutes after initiation of one-lung ventilation (OLV), (T3) 60 minutes after initiation of OLV, and (T4) 20 minutes after the end of OLV.
  Evaluation of Change in Peak inspiratory pressure (PIP).
Change in the MAP | four time points: (T1) 10 minutes after initiation of total lung ventilation (TLV), (T2) 10 minutes after initiation of one-lung ventilation (OLV), (T3) 60 minutes after initiation of OLV, and (T4) 20 minutes after the end of OLV.
  Evaluation of Change in Mean arterial pressure (MAP).
Change in the HR | four time points: (T1) 10 minutes after initiation of total lung ventilation (TLV), (T2) 10 minutes after initiation of one-lung ventilation (OLV), (T3) 60 minutes after initiation of OLV, and (T4) 20 minutes after the end of OLV.
  Evaluation of Change in Heart Rate (HR).

CONTACTS AND LOCATIONS:
Overall Officials: Faten Rostom, PHD, Study Chair — Department of Anesthesiology Faculty of Medicine Damascus University
Locations (1):
- University Children's Hospital, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Licker M, Hagerman A, Jeleff A, Schorer R, Ellenberger C. The hypoxic pulmonary vasoconstriction: From physiology to clinical application in thoracic surgery. Saudi J Anaesth. 2021 Jul-Sep;15(3):250-263. doi: 10.4103/sja.sja_1216_20. Epub 2021 Jun 19. PMID 34764832
- [Background] Kim D, Lee C, Bae H, Kim J, Oh EJ, Jeong JS. Comparison of the perfusion index as an index of noxious stimulation in monitored anesthesia care of propofol/remifentanil and propofol/dexmedetomidine: a prospective, randomized, case-control, observational study. BMC Anesthesiol. 2023 May 26;23(1):183. doi: 10.1186/s12871-023-02116-x. PMID 37237353
- [Background] Mahmoud M, Barbi E, Mason KP. Dexmedetomidine: What's New for Pediatrics? A Narrative Review. J Clin Med. 2020 Aug 24;9(9):2724. doi: 10.3390/jcm9092724. PMID 32846947
- [Background] De Cassai A, Boscolo A, Geraldini F, Zarantonello F, Pettenuzzo T, Pasin L, Iuzzolino M, Rossini N, Pesenti E, Zecchino G, Sella N, Munari M, Navalesi P. Effect of dexmedetomidine on hemodynamic responses to tracheal intubation: A meta-analysis with meta-regression and trial sequential analysis. J Clin Anesth. 2021 Sep;72:110287. doi: 10.1016/j.jclinane.2021.110287. Epub 2021 Apr 16. PMID 33873003
- [Background] Khddam A, Rostom F, Hajeer MY. Effect of Dexmedetomidine on Oxygen and Intrapulmonary Shunt (Qs/Qt) During One-Lung Ventilation in Pediatric Surgery: A Randomized Controlled Trial. Cureus. 2024 Mar 22;16(3):e56693. doi: 10.7759/cureus.56693. eCollection 2024 Mar. PMID 38523877
- [Background] Wang Y, Gong C, Yu F, Zhang Q. Effect of dexmedetomidine on intrapulmonary shunt in patients with sevoflurane maintained during one-lung ventilation: A case-control study. Medicine (Baltimore). 2022 Nov 18;101(46):e31818. doi: 10.1097/MD.0000000000031818. PMID 36401465
- [Background] Asri S, Hosseinzadeh H, Eydi M, Marahem M, Dehghani A, Soleimanpour H. Effect of Dexmedetomidine Combined with Inhalation of Isoflurane on Oxygenation Following One-Lung Ventilation in Thoracic Surgery. Anesth Pain Med. 2020 Feb 12;10(1):e95287. doi: 10.5812/aapm.95287. eCollection 2020 Feb. PMID 32309196
- [Background] Xu B, Gao H, Li D, Hu C, Yang J. Nebulized dexmedetomidine improves pulmonary shunt and lung mechanics during one-lung ventilation: a randomized clinical controlled trial. PeerJ. 2020 Jun 5;8:e9247. doi: 10.7717/peerj.9247. eCollection 2020. PMID 32547872
- [Background] Jiang H, Kang Y, Ge C, Zhang Z, Xie Y. One-lung ventilation patients: Clinical context of administration of different doses of dexmedetomidine. J Med Biochem. 2022 Apr 8;41(2):230-237. doi: 10.5937/jomb0-33870. PMID 35510198